CLINICAL TRIAL: NCT01098435
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Pilot Study of the Safety and Efficacy of RDC-0313 in Adults With Binge Eating Disorder
Brief Title: ALK33-101: A Study of RDC-0313 (ALKS 33) in Adults With Binge Eating Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK33-101
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Binge Eating Disorder
Keywords: Binge eating disorder; RDC-0313
MeSH Terms: conditions — Binge-Eating Disorder | interventions — ALKS-33

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RDC-0313 (ALKS 33) (Experimental): 2-capsules taken orally
  Interventions: Drug: RDC-0313 (ALKS 33)
- Placebo (Placebo Comparator): 2-capsules taken orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RDC-0313 (ALKS 33) — Capsules for daily oral administration
  Arms: RDC-0313 (ALKS 33)
Drug: Placebo — Capsules containing lactose and no active drug for daily oral administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety of daily doses of RDC-0313 (ALKS 33) compared with placebo in adults with binge-eating disorder (BED). An additional objective is to explore the efficacy of RDC-0313 treatment in comparison with placebo in adults with binge-eating disorder.

DETAILED DESCRIPTION:
Following screening, eligible subjects will be randomized in a 1:1 ratio to RDC-0313 (ALKS 33) or matching placebo. Once-daily at-home dosing will begin at randomization and will continue for 6 weeks. There will be 8 study visits over a 12-week study period. On an ongoing basis, subjects will complete a take-home binge diary designed to record the number of binge-eating episodes (binge episodes) and binge-eating days (binge days, days during which at least 1 binge occurred), as well as snacks and meals consumed daily over each 7-day period.

ELIGIBILITY:
Inclusion Criteria:

* Meet the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, text revised (DSM-IV-TR) criteria for a diagnosis of binge eating disorder (BED)
* Display greater than or equal to 3 binge eating days per week
* Body mass index (BMI) greater than or equal to 30 kg/m2
* Age of 18 years or older
* Women of childbearing potential must agree to use an approved method of birth control for the duration of the study

Exclusion Criteria:

* Concurrent symptoms of bulimia nervosa or anorexia nervosa
* Suicidal ideation
* DSM-IV-TR diagnosis of substance abuse or dependence (except nicotine or caffeine) within 6 months prior to randomization
* Positive urine toxicological screen for benzodiazepines, opioids, amphetamine/methamphetamine, or cocaine at screening or randomization
* Women who are pregnant or breastfeeding
* Participation in a psychological or weight loss intervention for BED that was initiated within the 3 months prior to screening
* Clinically unstable medical disease
* History of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* History of seizures, including clinically significant febrile seizures in childhood
* Current or anticipated need for prescribed opioid medication during the study period
* Use of any psychotropic medications (other than hypnotics)
* Participation in a clinical trial of a pharmacological agent within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Number of participants in each dose group reporting at least 1 treatment-emergent adverse event (TEAE) | 6 Weeks
  A TEAE is any adverse event (AE), regardless of causality, that either: begins after a participant's first dose of study drug, up to and including the final follow-up visit; or started before a participant's first dose of study drug but worsens in severity after the first dose of study drug, up to and including the final follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Marc deSomer, MD, Study Director — Alkermes, Inc.
Locations (6):
- United States (6):
  - Alkermes' Investigational Study Site, Tucson, Arizona
  - Alkermes' Investigational Study Site, Minneapolis, Minnesota
  - Alkermes' Investigational Study Site, Manlius, New York
  - Alkermes' Investigational Study Site, Raleigh, North Carolina
  - Alkermes' Investigational Study Site, Mason, Ohio
  - Alkermes' Investigational Study Site, Toledo, Ohio

REFERENCES:
- [Derived] McElroy SL, Guerdjikova AI, Blom TJ, Crow SJ, Memisoglu A, Silverman BL, Ehrich EW. A placebo-controlled pilot study of the novel opioid receptor antagonist ALKS-33 in binge eating disorder. Int J Eat Disord. 2013 Apr;46(3):239-45. doi: 10.1002/eat.22114. Epub 2013 Feb 5. PMID 23381803